CLINICAL TRIAL: NCT01248338
Title: Comparison the Effects of Nebivolol Versus Metoprolol Succinate on Endothelial Function and Large Artery Stiffness
Brief Title: Effects of Nebivolol Versus Metoprolol Succinate on Endothelial Function
Acronym: NEMENDAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Berlin-Chemie AG Menarini Group (Industry)
Responsible Party: Kaltwasser, Maria Theresia, Dr., Berlin-Chemie AG Menarini Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MeES/05/Neb-EnD/001
Record Dates: First submitted 2010-11-19; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Nebivolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- metoprolol, tablets (Active Comparator): metoprolol succinate 50-100 mg orally daily for one year
  Interventions: Drug: metoprolol succinate
- nebivolol (Experimental): nebivolol 5 mg capsule once daily for one year
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: metoprolol succinate — once daily 50 or 100 mg for one year
  Other Names: Corvitol
  Arms: metoprolol, tablets
Drug: Nebivolol — once daily 5 mg capsule for one year
  Other Names: Nebilet
  Arms: nebivolol

SUMMARY:
An impairment of endothelial function plays the central role in the pathogenesis of cardiovascular diseases and their complications. Most of cardiovascular risk factors are known to impair endothelial function and the established disease further aggravates endothelial dysfunction.

The aim of the present study is to investigate the effects of nebivolol or metoprolol succinate on endothelial function and large artery stiffness.

DETAILED DESCRIPTION:
The aim of this study was to compare the effects between the vasodilating β-blocker nebivolol and the cardioselective β-blocker metoprolol succinate on aortic blood pressure and left ventricular wall thickness. We conducted a randomized, double-blind study in 80 hypertensive patients. Patients received either nebivolol 5 mg or metoprolol succinate 50-100 mg daily for one year. Their heart rate, central and brachial blood pressure, mean arterial pressure, augmentation index, carotid-femoral pulse wave velocity and left ventricular wall thickness were measured at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate essential hypertension (systolic BP 140-179 mmHg and/or diastolic BP 90-109 mmHg)*
* Male and female patients aged 30-65 years Newly diagnosed untreated patients or previously diagnosed patients who were without treatment at least two weeks prior to screening* If patient has been taken previously antihypertensive medication the BP values are originated after untreated two weeks before randomization

Exclusion Criteria:

* Concomitant medication: Cyclic antidepressants, MAO inhibitors, corticosteroids
* Diabetes I or II type (fasting venous plasma glucose > 6.4 mmol/l)
* Bronchial asthma and chronic obstructive airway disease
* Body mass index > 30 kg/m2
* Ischaemic heart disease (III, IV stage, Canadian Cardiovascular Society)
* Clinically relevant heart failure (NYHA class II - IV)
* Clinically relevant valve disease (physical examination)
* Arrhythmias and conduction disturbances, requiring therapy, sinus bradycardia at rest < 50 b/min, sick sinus syndrome, AV - block stage II - III
* Secondary hypertension (urea >8.3 mmol/l, creatinine >120μmol/l (males), >103 μmol/l (females), TSH > 4.0mIU/l, free T4 > 27 pmol/l)
* Clinically relevant atherosclerotic disease of lower extremities
* Acute inflammation (according to CRP > 10mg/l)
* Hypercholesterolemia (> 6,5 mmol/l)
* Allergic reaction to beta-blockers
* Pregnant or breast-feeding women
* History of hepatic, renal, metabolic or endocrine diseases
* Smoking > 10 cigarettes per day
* Alcohol consumption > 7 drinks per week (drink = 0,33 l beer, 120 ml wine or 30 ml strong alcoholic drink)
* The patient has had surgery or disease of the gastrointestinal tract which, in the opinion of the investigator, may influence the absorption or elimination of the study drug.
* The patient has a severe organic disorder that may interfere with the absorption, pharmacokinetics, or elimination of the study medication.
* The patient has a comorbid condition that would be expected to result in death during the trial period (e.g., terminal cancer, AIDS).
* The patient has chronic psychoses or behavioural conditions that would limit the ability of the patient to comply with the requirements of this study.
* The patient has known hypersensitivity to Nebivolol, Metoprolol or hydrochlorothiazide related compounds.
* Patient is enrolled in another clinical trial.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Effects of nebivolol and metoprolol on endothelial function | 12 months
  High-fidelity micromanometer (applanation tonometry) from both wrists and PWA, which is to be performed of the systolic portion (SphygmoCor Px, version 7.0) of the pulse curve.

SECONDARY OUTCOMES:
Change in carotid artery intima-media thickness | 12 months
  Ultrasound scanner,with an 12 MHz transducer. Longitudinal images from 3 projections (anterolateral, lateral, and posterolateral) are measured for the common carotid artery, carotid bulb, and internal carotid artery
Change in left ventricular mass index, systolic and diastolic function | 12 months
  2-dimensional echocardiography using the standard apical 4-chamber view
Arterial Compliance | 12 months
  Peripheral blood pressure and arterial waveform to be measured in the dominant arm by a Cardiovascular Profiling Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Jaan Eha, Professor, Principal Investigator — Cardiology Clinic of Tartu University Clinics
Locations (1):
- Cardiology Clinic of Tartu University Clinics, Tartu, Estonia, Estonia

REFERENCES:
- [Derived] Serg M, Kampus P, Kals J, Zagura M, Zilmer M, Zilmer K, Kullisaar T, Eha J. Nebivolol and metoprolol: long-term effects on inflammation and oxidative stress in essential hypertension. Scand J Clin Lab Invest. 2012 Sep;72(5):427-32. doi: 10.3109/00365513.2012.691991. Epub 2012 Jun 18. PMID 22708640
- [Derived] Kampus P, Serg M, Kals J, Zagura M, Muda P, Karu K, Zilmer M, Eha J. Differential effects of nebivolol and metoprolol on central aortic pressure and left ventricular wall thickness. Hypertension. 2011 Jun;57(6):1122-8. doi: 10.1161/HYPERTENSIONAHA.110.155507. Epub 2011 May 2. PMID 21536983